CLINICAL TRIAL: NCT06845345
Title: Effect of Mediterranean Diet Combined With Intermittent Fastingon Liver Fibrosis Compared to Naltrexone/Bupropion in People With Cardiometabolic Risk Factors
Brief Title: Effect of Mediterranean Diet Combined With Intermittent Fasting on Liver Fibrosis Compared to Naltrexone/Bupropion in People With Cardiometabolic Risk Factors (MEDFAST-study)
Acronym: MEDFAST
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Carmen Dietvorst (Other)
Responsible Party: Sponsor-Investigator, Carmen Dietvorst, MSc., Franciscus Gasthuis
Organization: Franciscus Gasthuis (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-519774-40-00; 2024-519774-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-17; First posted 2025-02-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2; Liver Fibrosis; Liver Steatoses; Hepatic Steatosis; Hepatic Fibrosis; Overweight or Obesity; MASLD; MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; Cardio-metabolic Risk; Cardio-metabolic Health; Hypertension; Dyslipidaemia
Keywords: diabetes; liver diseases; liver fibrosis; intermittent fasting; mediterranean diet; mysimba; lifestyle; cardiometabolic diseases; obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Liver Cirrhosis; Fatty Liver; Overweight; Obesity; Hypertension; Dyslipidemias; Diabetes Mellitus; Liver Diseases; Intermittent Fasting | interventions — Diet, Mediterranean; Diet Therapy; bupropion hydrochloride, naltrexone hydrochoride drug combination; Naltrexone; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary arm (Active Comparator): Calorie restricted Mediterranean diet, with an eating window between 8AM till 6PM (early time-restricted eating)
  Interventions: Other: early time restricted Mediterranean diet
- Pharmacological arm (Active Comparator): 32 mg/360 mg naltrexone/bupropion (Mysimba)
  Interventions: Drug: Mysimba

INTERVENTIONS:
Other: early time restricted Mediterranean diet — Participants will start with a calorie restricted Mediterranean diet, with an eating window between 8AM till 6PM (early time-restricted eating) for a period of six months. Participants are asked to stop eating at 6PM. This results in a daily fasting window of approximately 14 hours. A daily caloric intake of 500 kcal compared to the calculated energy requirement is assumed to stimulate weight loss.
  Other Names: early time restricted eating; mediterranean diet; intermittent fasting; dietary intervention
  Arms: Dietary arm
Drug: Mysimba — Participants will take Mysimba twice daily at a total dose of 32 mg/360 mg naltrexone/bupropion per day for a duration of six months. The dosage will be built up in the first month following the stepped care approach used in the SmPC. Participants receive usual care, including the advice of 60 minutes of exercise per day and standard dietary recommendations according to the guidelines for the Dutch population.
  Other Names: naltrexone/bupropion; pharmacological intervention
  Arms: Pharmacological arm

SUMMARY:
In the Netherlands, there are many people with cardiometabolic diseases. More than half of these people also have fatty liver. This is a build-up of fat in the liver (steatosis) and can lead to long-term scarring (fibrosis) and even death of the liver. Losing weight can help reduce this. Losing weight can be done with medication such as naltrexone/bupropion (Mysimba®), which is often prescribed to people with cardiometabolic diseases, but losing weight can also be done with diet. In this study, the investigators want to combine a Mediterranean diet (with lots of vegetables, fruits, whole grain products, nuts and olive oil) with intermittent fasting. In addition participants are not allowed to eat after the evening meal. The investigators will compare this with a group of participants receiving Mysimba®, to see if a diet with intermittent fasting might be better for reducing liver steatosis and fibrosis in people with cardiometabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 27 kg/m2 and at least one cardiometabolic risk factor (type 2 diabetes, hypertension, dyslipidaemia) or BMI > 30
* Moderate to severe liver fibrosis (LSM >7.0 kPa and <13.6 kPa)
* Aged 18-75 years
* Written informed consent

Exclusion Criteria:

* An insufficient comprehension of the Dutch language (spoken and written)
* Female who is pregnant, breast-feeding or intends to become pregnant
* Participants with an established diagnosis of liver pathology like, but not limited to: Hepatitis B, Hepatitis C, Autoimmune hepatitis, Wilson's disease, Hemochromatosis, Primary biliary cholangitis, Primary sclerosing cholangitis, Alcoholic liver disease
* History of liver transplant, or current placement on a liver transplant list
* History of cirrhosis and/or hepatic decompensation, including ascites, hepatic encephalopathy or variceal bleeding
* Participants with active HIV infection and/or treatment
* Participants with diagnosed malignancies with or without active treatment
* Participants with history or pre-existing renal disease (eGFR <30 mL/min/1.73 m2)
* Participants with corticosteroid induced diabetes (while still using corticosteroids)
* Participants using GLP-1 agonists for less than 3 months or not yet on a stable dose
* Participants using MAO-inhibitors, opioids and/or methadone (due to contraindication)
* Known or suspected excessive alcohol consumption (>21 drinks/week for males or >14 drinks/week for females. One drink is equivalent to 10 grams of alcohol)
* Previous or planned (during the trial period) obesity treatment with surgery. However, previous interventions that, due to reversal or removal, do not have any influence on the patient's weight, in the opinion of the investigator, are allowed.
* Participants with a history or evidence of any other clinically significant condition or planned or expected procedure that in the opinion of the investigator, may compromise the patient's safety or ability to complete the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender men and women
Enrollment: 70 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Between-group difference in liver fibrosis during six months | Change from baseline to 6 months
  Measured as liver stiffness in kilopascals (kPa) by transient elastography with FibroScan. For a value between 0 and 8 kPa, no liver fibrosis is assumed. Anything above 8 kPa means liver fibrosis. The highest possible result is 75 kPa.

SECONDARY OUTCOMES:
Between group difference in liver steatosis during six months | Change from baseline to 6 months
  Measured as Controlled Attenuation Parameter (CAP) score with FibroScan. This score will range from 100 to 400 decibels per meter (dB/m). A score below 238 dB/m means the amount of fatty change in the liver is not higher than normal.
Between-group difference in weight during six months | Change from baseline to 6 months
  Measured in kilograms (kg) with Seca 888 compact digital flat scale. Along with height, BMI is calculated by dividing weight by height squared. BMI should be at least 27 kg/m^2.
Between-group difference in height during six months | Change from baseline to 6 months
  Measured in centimeters (cm) with a yardstick. Along with weight, BMI is calculated by dividing weight by height squared. BMI should be at least 27 kg/m^2.
Between-group difference in waist circumference during six months | Change from baseline to 6 months
  Measured in centimeters (cm) with measuring tape. A healthy waist circumference for women is between 68 and 80 cm and for men between 79 and 94 cm.
Between-group difference in body composition during six months | Change from baseline to 6 months
  Impedance, resistance and reactance are measured in Ohm at 50 kHz with bioelectrical impedance analysis (Bodystat 500). The impedance measuring range is between 20 and 1300 Ohm.
Between-group difference in grip strength during six months | Change from baseline to 6 months
  Measured in kilograms (kg) with a hand dynamometer (Jamar). The grip strength can be measured between 0 and 90 kg. Normal values depend on gender and age. In people aged 20-29, the average grip strength is 46 kg for men and 29 kg for women.
Between-group difference in glycaemic regulation during six months | Change from baseline to 6 months
  Glycaemic regulation is determined from values measured in the blood. These include fasting blood glucose measured in millimoles per litre (mmol/l), haemoglobin A1c (HbA1c) measured in millimoles per mole (mmol/mol) and fasting insulin measured in milligrams per decilitre (mg/dl). Normal values are below 6.1 mmol/l for fasting glucose, below 53 mmol/mol for HbA1c and between 60-110 mg/dl for fasting insulin.
Between-group differences in cholesterol during six months | Change from baseline to 6 months
  Total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides are measured in millimoles per litre (mmol/l) through blood samples. Normal values are <5.0 mmol/l for total cholesterol, <2.6 for LDL cholesterol, >0.8 for HDL cholesterol and <2.0 for triglycerides
Between-group differences in lipoproteins during six months | Change from baseline to 6 months
  Apolipoprotein B (ApoB), apolipoprotein AI (ApoAI), lipoprotein a (Lp(a)) and Apolipoproteïne B48 are measured in grams per litre (g/l) through blood samples. Normal values are: ApoB 0.55-1.4 g/l for men and 0.55-1.25 g/l for women; ApoAI 1.1-2.05 g/l for men and 1.25-2.15 g/l for women; Lp(a) <0.5 g/l. There are no normal values for Apolipoprotein B48 yet.
Between-group difference in blood pressure during six months | Change from baseline to 6 months
  Systolic and diastolic blood pressure measured in millimetres of mercury pressure (mmHg). Normal values are 120-140 mmHg for systolic pressure and <90 mmHg for diastolic pressure.
Between-group difference in liver enzymes during six months | Change from baseline to 6 months
  Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are measured in units per litre (U/L). Normal values are <50 U/L for men and <35 U/L for women for ALT and <40 U/L for men and <32 U/L for women for AST.
Between-group difference in renal function during six months | Change from baseline to 6 months
  Renal function is determined by measuring creatinine in micromol per litre (µmol/L) and eGFR in mL/min/1.73m^2. Normal values are 62-106 µmol/L for men and 44-80 µmol/L for women for creatinine; >90 mL/min/1.73m^2 for eGFR.
Between-group difference in blood count during six months | Change from baseline to 6 months
  Blood count is determined by thrombocytes and leukocytes in x10⁹/L. Normal values are 150-400 x10⁹/L for thrombocytes and 4.0-10.0 x10⁹/L for leukocytes.
Between-group difference in physical activity during six months | Change from baseline to 6 months
  Physical activity will be measured with Activ8 Activity Tracker GEN2. Activity is measured in time (seconds), Metabolic equivalent (MET) and kilocalories (kcal). All for sitting, standing, walking, cycling, running and total/average. In addition, step count is also measured.
Between-group difference in lifestyle factors during six months | Change from baseline to 6 months
  Food intake, demographic variables, drug use, smoking and drinking habits, (diabetes) medication use and compliance to the time restriction will be administered with a self-developed questionnaire
Between-group difference in quality of life during six months | Change from baseline to 6 months
  Measured with SF-36 Questionnaire. This is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a total higher score defining a more favorable health state.
Between-group difference in patient satisfaction during six months | Change from baseline to 6 months
  Measured with Diabetes Treatment Satisfaction Questionnaire. It consists of 8 items, indicating how satisfied a person is with diabetes treatment. The score can be a minimum of 0 and a maximum of 36. The higher the score the more satisfied.

OTHER OUTCOMES:
Shift in liver fibrosis severity during six months | Change from baseline to 6 months
  Liver fibrosis is categorized in fibrosis score F0, F1, F2 or F3. The scores are classified according to liver stiffness (kPa). Fibrosis score F0 and F1 means normal (no scarring), F2 means moderate scarring and F3 means severe scarring. The lower the score the better.
Drop-outs during six months | Change from baseline to 6 months
  Number of participants that drop-out (categorized by reason for drop-out)
Side effects during six months | Change from baseline to 6 months
  Side effects will be self-reported

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Castro Cabezas, Dr., Principal Investigator — Franciscus
Locations (1):
- Franciscus, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
All individual data will be encrypted and shared only with the research team.